CLINICAL TRIAL: NCT01198834
Title: A Randomized, Multi-Center, Double-Blind, Factorial, Comparator and Placebo-Controlled Phase III Trial to Evaluate the Efficacy, Tolerability and Safety of MRX-7EAT Etodolac-Lidocaine Topical Patch in the Treatment of Ankle Sprains
Brief Title: MRX-7EAT Etodolac-Lidocaine Topical Patch in the Treatment of Ankle Sprains
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: MEDRx USA, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: MRX-7EAT-1005
Record Dates: First submitted 2010-09-09; First posted 2010-09-10 (Estimated); Last update posted 2018-01-17 (Actual); Status verified 2018-01

CONDITIONS: Ankle Sprains
Keywords: ankle sprains
MeSH Terms: conditions — Ankle Injuries | interventions — Lidocaine; Etodolac

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Placebo Patch (Placebo Comparator): Treatment with Placebo Patch
  Interventions: Drug: Placebo
- MRX-7EAT Patch (Experimental): Treatment with MRX-7EAT Patch
  Interventions: Drug: MRX-7EAT
- Lidocaine Patch (Experimental): Treatment with Lidocaine Patch
  Interventions: Drug: Lidocaine
- Etodolac Patch (Experimental): Treatment with Etodolac Patch
  Interventions: Drug: Etodolac

INTERVENTIONS:
Drug: MRX-7EAT — Application of up to two patches at the discretion of the investigator for up to 7 days.
  Arms: MRX-7EAT Patch
Drug: Placebo — Application of up to two patches at the discretion of the investigator for up to 7 days.
  Arms: Placebo Patch
Drug: Lidocaine — Application of up to two patches at the discretion of the investigator for up to 7 days.
  Arms: Lidocaine Patch
Drug: Etodolac — Application of up to two patches at the discretion of the investigator for up to 7 days.
  Arms: Etodolac Patch

SUMMARY:
A Randomized, Multi-Center, Double-Blind, Factorial, Comparator and Placebo-Controlled Phase III Trial to Evaluate the Efficacy, Tolerability and Safety of MRX-7EAT Etodolac-Lidocaine Topical Patch in the Treatment of Ankle Sprains

ELIGIBILITY:
Inclusion Criteria

A subject will be eligible for inclusion in this study if all of the following criteria apply:

1. Subject has signed an informed consent form.
2. Subject is 14 years of age or older (with assent according to state law).
3. Females of child bearing potential must have a negative pregnancy test and be using an adequate method of birth control. Adequate is defined as either hormonal or partner vasectomy for at least three months, or , condoms, IUD, abstinence or other prescribed birth control. Females may be considered non-childbearing if post-menopausal at least 1 year or surgically sterile.
4. Subject has a diagnosis of uncomplicated acute soft tissue inversion injury of the ankle, Grade II classification (as defined by the American Academy of Orthopaedic Surgeons (AAOS), "partial tearing of the ligament") that has occurred ≥ 6 hours to ≤ 48 hours before study entry.
5. Subject has a Current Pain Intensity during point and flex with the ankle unwrapped rated prior to study entry as ≥ 5 but ≤ 8 on an NPRS (11 point; range 0 to 10; anchors to be "none" and "severe").
6. Subject is willing and able to comply with the protocol.

Exclusion Criteria

A subject will not be eligible for inclusion in this study if any of the following criteria apply:

1. Females of child bearing potential that are not using an adequate method of birth control or are breastfeeding (adequate defined as either hormonal or partner vasectomy for at least three months, or other prescribed birth control, condoms, IUD, abstinence or other prescribed birth control).
2. Subject has a Grade I ("slight stretching and some damage to the fibers (fibrils) of the ligament") or Grade III ("complete tear of the ligament") sprain or strain, bilateral sprain or strain, or concomitant fracture or open wound at the site of the sprain or strain, or has a serious injury, as determined by the investigator (e.g., nerve damage, joint instability, or tendon rupture); or surgical treatment is required. Diagnosis of Grade III is indicated by a positive anterior drawer test or positive talar tilt test is exclusionary (inability to perform test(s) is exclusionary when in the opinion of the investigator a Grade III sprain is suspected).
3. Subject has a history of a previous injury to the same area within two months prior to current injury or previous surgery in the same area.
4. Subject has used non-pharmacologic treatments for the injury within 2 hours prior to the baseline visit (e.g. ice or acupuncture) that may interfere with pain assessments. Subjects on any therapeutic exercise regimen should continue based on the investigator's discretion. Use of iontophoresis is prohibited.
5. Subject has used oral pharmacologic treatments (NSAIDs or analgesic medications) for the injury less than three half-lives before the baseline assessments; ibuprofen is permitted prior to baseline as long as it is not within six hours of the baseline assessment aspirin (81-325 mg daily) taken prophylactically for cardiovascular reasons is permitted.
6. Subject has used any form of opioid within 24 hours of study entry or used opioids for five or more consecutive days within the 30 days preceding the screening visit.
7. Subject has received systemic corticosteroids in the 30 days preceding the screening visit (e.g., intra-articular, peritendinous, oral, or parenteral administration); topical corticosteroid use is acceptable unless applied to the target joint; and inhaled steroids are acceptable (e.g. Flonase®).
8. Subject recently initiated sleep medications, muscle relaxants, anticonvulsants or antidepressants (within the past 30 days); if using any of these, subject must be on a stable dose and regimen for 30 days prior to study enrollment.
9. Subject has used TNF alpha blockers or Class 1 anti-arrhythmic drugs within the 60 days preceding the screening visit.
10. Subject has a history or physical assessment finding of clinically significant GI ulcers or abnormal bleeding, anemia, kidney disease, liver disease, poorly controlled lung, stomach, heart, or other vital organ disease as determined by the study investigator/physician.
11. Subject has a history or physical assessment finding that is not compatible with safe participation in the study as determined by the study investigator.
12. Subject has any form of inflammatory arthritis, spondyloarthropathies (sPA), fibromyalgia, or is currently undergoing treatment for chronic pain; or has a history of, or evidence for, underlying disease in the injured area, such as osteoarthritis or gout.
13. Subject has any pain or medical problem that, in the investigator's opinion, may interfere with pain measurement of the target joint.
14. Subject has active skin lesions or disease at the intended site of application of the study medication. Skin lesions include open wounds, rash, papules and vesicles; abrasions, lacerations or any break in skin at the intended site of patch application.
15. Subject has a history of allergy to etodolac, other NSAIDs, lidocaine, or adhesives (e.g. adhesive tape).
16. Subject has a history of prior failed treatment with topical NSAIDs (Flector® Patch or Voltaren® Gel) defined as repeated attempts within the three months preceding the screening visit.
17. Subject has a history of drug or alcohol abuse within the past two years preceding the screening visit.
18. Subject has received an investigational drug or product or participated in an investigational drug study within a period of 30 days prior to receiving study medication.
19. Subject has scheduled elective surgery or other invasive procedures during the period of study participation.
20. Subject is on workman's compensation or has pending legal hearings associated with any injury.
21. Subject refuses to provide informed consent or is unwilling or unable to follow study procedures.

Min Age: 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 600 (Actual)
Dates: Start 2010-09; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Mean of All Current Pain Intensity During Point and Flex Scores on Days 2 Through 7 on a 0-10 Numeric Pain Rating Scale (NPRS). | Days 2 to 7

SECONDARY OUTCOMES:
Current Pain Intensity during Point and Flex | Days 1 through 7
Current Pain Intensity at Rest, Passive Stretch and Pain Intensity While Standing On a Single Foot | Each Clinical Visit
Impact on Physical Function | Days 1 to 7
Total Number of Patches Used | Days 1 to 7
Time to Pain Resolution | Days 1 to 7
Assessment of Patch Adherence | Clinical Visit 2
Subject's Treatment Satisfaction | Clinical Visit 3

CONTACTS AND LOCATIONS:
Overall Officials: Martine Francis, Study Director — IL Pharma
Locations (33):
- United States (33):
  - Phoenix, Arizona
  - North Little Rock, Arkansas
  - Chico, California
  - Palm Springs, California
  - San Diego, California
  - Aurora, Colorado
  - Colorado Springs, Colorado
  - Denver, Colorado
  - Daytona Beach, Florida
  - Fort Lauderdale, Florida
  - Gulf Breeze, Florida
  - Orlando, Florida
  - West Palm Beach, Florida
  - Boise, Idaho
  - Avon, Indiana
  - Fishers, Indiana
  - Franklin, Indiana
  - Greenfield, Indiana
  - Muncie, Indiana
  - Dubuque, Iowa
  - Wichita, Kansas
  - Erlanger, Kentucky
  - Henderson, Nevada
  - Charlotte, North Carolina
  - Fargo, North Dakota
  - Cincinnati, Ohio
  - Oklahoma City, Oklahoma
  - Georgetown, Texas
  - Lubbock, Texas
  - San Antonio, Texas
  - Temple, Texas
  - Riverton, Utah
  - Danville, Virginia